CLINICAL TRIAL: NCT07375966
Title: Repeated Intravenous Thrombolysis for Ischemic Stroke With Medium to Large Vessel Occlusion Presenting Within 4.5 Hours of Onset With Tenecteplase (RITIS-TNK2): a Prospective, Randomized, Open Label, Blinded Assessment of Outcome, and Multi-center Study
Brief Title: Repeated Intravenous Thrombolysis for Ischemic Stroke With Medium to Large Vessel Occlusion Presenting Within 4.5 Hours of Onset With Tenecteplase (RITIS-TNK2)
Acronym: RITIS-TNK2
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: General Hospital of Shenyang Military Region (Other)
Responsible Party: Principal Investigator, Hui-Sheng Chen, Director, General Hospital of Shenyang Military Region
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Y (2025) 502
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Ischemic Stroke
MeSH Terms: conditions — Ischemic Stroke | interventions — Tenecteplase

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TNK group (Experimental): Tenecteplase is administered intravenously at a dose of 16 mg, with a maximum dose of 0.25 mg/kg.
  Interventions: Drug: Tenecteplase
- Control group (No Intervention): no tenecteplase

INTERVENTIONS:
Drug: Tenecteplase — Tenecteplase is administered intravenously at a dose of 16 mg, with a maximum dose of 0.25 mg/kg.
  Arms: TNK group

SUMMARY:
While intravenous thrombolysis (IVT) within 4.5 hours is the standard medical reperfusion therapy, its efficacy is limited, particularly for large or medium vessel occlusions (LVO/MeVO), with low recanalization rates for IVT with rt-PA. The newer thrombolytic agent, tenecteplase (TNK), offers practical advantages-including single bolus administration, a longer half-life, and potentially higher fibrin specificity-and has been shown to be non-inferior to rt-PA.

Despite advances, a significant proportion of patients with LVO/MeVO do not achieve early clinical improvement after standard IVT, likely due to persistent occlusion from a high thrombus burden. Endovascular therapy, while highly effective for LVO, has limited accessibility. Therefore, there is an urgent need for more effective and widely accessible pharmacological strategies.

This study proposes a rescue strategy based on the hypothesis that a second dose of IVT may improve outcomes in patients with imaging-confirmed LVO or MeVO who show no significant neurological improvement one hour after standard TNK thrombolysis (administered within 4.5 hours of stroke onset). The primary aim of this study is to formally evaluate the efficacy and safety of a repeated dose of intravenous tenecteplase in this specific patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 year;
* Acute ischemic stroke presumably caused by large or medium vessel occlusion within 4.5 hours of onset, having received standard-dose intravenous thrombolysis, and with no planned thrombectomy;
* Measurable neurological deficit before the first intravenous thrombolysis, with NIHSS ≥ 4;
* Baseline pc-ASPECTS/ASPECTS ≥ 6, and for posterior circulation infarction, a Pontine-Midbrain Index ≤ 2 (assessed by CT or DWI);
* No significant clinical improvement (reduction in NIHSS ≤ 2) or neurological deterioration after initial improvement at 1 hour after the first thrombolysis;
* Follow-up imaging (CTA or MRA) at 1 hour after the first thrombolysis rules out intracranial hemorrhage and confirms the presence of large or medium vessel occlusion (internal carotid artery, M1-M3 segments of the middle cerebral artery, A1-A3 segments of the anterior cerebral artery, P1-P3 segments of the posterior cerebral artery, basilar artery or V4 segment of the vertebral artery, PICA, AICA, or SCA);
* The second intravenous thrombolysis can be administered within 6 hours of onset;
* First stroke onset or past stroke without obvious neurological deficit (mRS≤1);
* Signed informed consent.

Exclusion Criteria:

* Planed for endovascular treatment;
* Significant white matter hyperintensities (Fazekas score 3);
* Any coagulation abnormality before the first thrombolysis, including INR > 1.5;
* Receipt of dual antiplatelet therapy within 24 hours prior to thrombolysis.；
* Pregnancy；
* Allergy to the investigational drug(s)；
* Comorbidity with other serious diseases;
* Participating in other clinical trials within 3 months;
* Patients not suitable for the study considered by researcher.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
rate of vessel recanalization | 24 (-6/+12) hours

SECONDARY OUTCOMES:
proportion of excellent functional outcome (modified Rankin Scale (mRS) 0-1) | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
proportion of favorable functional outcome (modified Rankin Scale (mRS) 0-2) | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
ordinal distribution of modified Rankin Scale (mRS) | 90±7 days
  The minimum and maximum values of mRS are 0 and 6, respectively; higher score mean a worse outcome
occurrence of early neurological improvement (ENI) | 24 (-6/+12) hours
  ENI is defined as more than 4-point decrease in National Institute of Health stroke scale score
change in National Institute of Health stroke scale (NIHSS) score | 24 (-6/+12) hours
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome
change in National Institute of Health stroke scale (NIHSS) score | 10±2 days
  the minimum and maximum values of NIHSS are 0 and 42, respectively; higher NIHSS mean a worse outcome
all-cause mortality | 10±2 days
occurence of symptomatic intracranial hemorrhage (sICH) | 24 (-6/+12) hours
occurence of any intracranial hemorrhage | 24 (-6/+12) hours
occurence of major systemic bleeding event | 24 (-6/+12) hours
occurence of any bleeding event | 24 (-6/+12) hours

CONTACTS AND LOCATIONS:
Locations (1):
- Lu Wang, Shenyang, Liaoning, China